CLINICAL TRIAL: NCT00422513
Title: A Randomized, Open-label Study Comparing the Pharmacoeconomic (Time and Motion) Benefit of Mircera and Epoetin Alfa in Patients With Chronic Kidney Disease (Stage V) on Dialysis.
Brief Title: A Study Comparing Mircera and Epoetin Alfa for the Treatment of Anemia in Dialysis Patients With Chronic Kidney Disease.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic decision unrelated to safety or efficacy
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20336
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator; Epoetin Alfa

ARMS (2):
- methoxy polyethylene glycol-epoetin beta (Experimental): 120-360 micrograms (iv) monthly, starting dose
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta
- Epoetin Alfa (Active Comparator): As prescribed, (iv), 3 times weekly
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta — 120-360 micrograms intravenous (iv) monthly, starting dose
  Other Names: Mircera
  Arms: methoxy polyethylene glycol-epoetin beta
Drug: Epoetin alfa — As prescribed, iv, 3 times weekly
  Arms: Epoetin Alfa

SUMMARY:
This 2 arm study will compare 'time and motion' (provider time spent on anemia management) and effect on hemoglobin (Hb) levels, of methoxy polyethylene glycol-epoetin beta (Mircera) and epoetin alfa, in anemic patients with chronic kidney disease (CKD) on hemodialysis. Patients stable on intravenous (iv) epoetin alfa will be randomized either to receive standard of care therapy (epoetin alfa (iv) 3 times weekly), or to receive Mircera 120-360 micrograms (iv), monthly. After a titration period, average time spent on anemia treatment over a 3 month period will be evaluated. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* CKD (stage V) on outpatient hemodialysis therapy for >= 3 months;
* CKD-related anemia treated with epoetin alfa iv 3x/week for >= 3 months;
* average hemoglobin (Hb) 10-12 g/dL over last 3 months.

Exclusion Criteria:

* failed renal transplant within 12 months prior to screening;
* poorly controlled hypertension;
* previous treatment with Mircera.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (44):
- United States (44):
  - Birmingham, Alabama
  - Rainbow City, Alabama
  - Hot Springs, Arizona
  - Fairfield, California
  - Los Alamitos, California
  - Los Angeles, California
  - Mountain View, California
  - Riverside, California
  - San Diego, California
  - Simi Valley, California
  - Whittier, California
  - Lakewood, Colorado
  - Brandon, Florida
  - Hudson, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Ocala, Florida
  - Palm Beach Gardens, Florida
  - Augusta, Georgia
  - Gurnee, Illinois
  - Fort Wayne, Indiana
  - Detroit, Michigan
  - Pontiac, Michigan
  - Sparks, Nevada
  - New Brunswick, New Jersey
  - Brooklyn, New York
  - Brooklyn Center, New York
  - Flushing, New York
  - Orchard Park, New York
  - The Bronx, New York
  - Williamsville, New York
  - Raleigh, North Carolina
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Lancaster, Pennsylvania
  - Lewistown, Pennsylvania
  - Philadelphia, Pennsylvania
  - West Homestead, Pennsylvania
  - Columbia, South Carolina
  - Orangeburg, South Carolina
  - Corpus Christi, Texas
  - Houston, Texas
  - Chesapeake, Virginia
  - Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa
Started | 130 | 130
Completed | 23 | 24
Not Completed | 107 | 106
Not completed — Lack of Efficacy | 4 | 5
Not completed — Protocol Violation | 23 | 7
Not completed — Refused Treatment | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — early termination of the study | 67 | 80
Not completed — Adverse Event | 4 | 4
Not completed — Death | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa | Total
Number analyzed (Participants) | 123 | 129 | 252
Age Continuous [Mean (Standard Deviation); unit: years] — Eight patients were excluded from the safety population: 7 patients in the Methoxy Polyethylene Glycol-epoetin Beta group and 1 patient in the epoetin alfa group. Six patients in the Methoxy Polyethylene Glycol-epoetin Beta group did not receive study medication. Seven patients in the Methoxy Polyethylene Glycol-epoetin Beta group and 1 patient in the epoetin alfa group did not have a postbaseline safety assessment.
  years | 59.3 (13.90) | 60.0 (14.06) | 59.7 (13.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 60 | 112
  Male | 71 | 69 | 140

OUTCOME MEASURES:

1. Primary Outcome: Time Spent on Anemia Treatment Over Evaluation Period
Description: Efficacy and pharmacoeconomics analyses were not performed.
Time Frame: Months 5-7
Population: The safety population was the anticipated population analyzed. Efficacy and pharmacoeconomics analyses were not performed.
Measure: Number; unit: months
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Hemoglobin (Hb) Concentration From Baseline to the Average Over the Evaluation Period
Description: Efficacy and pharmacoeconomics analyses were not performed.
Time Frame: Baseline, Months 5-7
Population: as for outcome 1
Measure: Number; unit: g/dL
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Assessed for AEs
Description: The adverse events are captured in the adverse event and serious adverse event section of this database.
Time Frame: Month 1 to 15 day follow up post month 7
Population: Safety Population
Measure: Number; unit: number of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa
Number analyzed (Participants) | 123 | 129
number of participants | 123 | 129

4. Secondary Outcome: The Number of Participants With Marked Laboratory Abnormalities Occurring in ≥5% of the Participants
Description: A marked laboratory abnormality was defined as a test result that was outside of the marked abnormality range and that also represented a clinically relevant change from baseline of at least a designated amount.
Time Frame: Baseline, Month 1 to Month 7
Population: Safety Population
Measure: Number; unit: number of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa
Number analyzed (Participants) | 123 | 129
number of participants
  Hematocrit - low | 32 | 24
  Hemoglobin - low | 36 | 28
  Platelets - low | 9 | 4
  Creatine Phosphokinase - high | 4 | 8
  Potassium - high | 20 | 20
  Fasting Glusose - high | 20 | 20
  Phosphate - high | 52 | 48
  Phosphate - low | 9 | 12

ADVERSE EVENTS:
Time Frame: Month 1 to 15 day follow up post month 7
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta | Epoetin Alfa
Serious Adverse Events (participants affected / at risk) | 24/123 | 38/129
Other Adverse Events (participants affected / at risk) | 15/123 | 21/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=123) | Epoetin Alfa (N=129)
cardiac failure congestive (Cardiac disorders) | 0 | 11
myocardial infarction (Cardiac disorders) | 0 | 3
coronary artery disease (Cardiac disorders) | 2 | 1
cardiac arrest (Cardiac disorders) | 1 | 1
acute coronary syndrome (Cardiac disorders) | 0 | 1
coronary artery occlusion (Cardiac disorders) | 1 | 0
sick sinus syndrome (Cardiac disorders) | 0 | 1
ventricular fibrillation (Cardiac disorders) | 1 | 0
pneumonia (Infections and infestations) | 1 | 3
arteriovenous graft site infection (Infections and infestations) | 2 | 0
bacterial sepsis (Infections and infestations) | 0 | 2
bronchitis (Infections and infestations) | 1 | 0
gastroenteritis (Infections and infestations) | 0 | 1
gastroenteritis viral (Infections and infestations) | 0 | 1
pseudomembranous colitis (Infections and infestations) | 1 | 0
pyelonephritis (Infections and infestations) | 1 | 0
vulval abscess (Infections and infestations) | 1 | 0
appendiccal mucocoele (Gastrointestinal disorders) | 1 | 0
colitis (Gastrointestinal disorders) | 0 | 1
colitis ischaemic (Gastrointestinal disorders) | 0 | 1
colonic pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
diabetic gastropathy (Gastrointestinal disorders) | 0 | 1
gastric ulcer (Gastrointestinal disorders) | 0 | 1
gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
intestinal obstruction (Gastrointestinal disorders) | 0 | 1
peptic ulcer (Gastrointestinal disorders) | 0 | 1
hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
fluid overload (Metabolism and nutrition disorders) | 0 | 1
hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 | 0
hypertension (Vascular disorders) | 1 | 2
malignant hypertension (Vascular disorders) | 1 | 0
peripheral vascular disorder (Vascular disorders) | 0 | 1
thrombosis (Vascular disorders) | 0 | 1
vascular calcification (Vascular disorders) | 1 | 0
vascular pseudoaneurysm ruptured (Vascular disorders) | 1 | 0
arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
hand fracture (Injury, poisoning and procedural complications) | 1 | 0
lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
overdose (Injury, poisoning and procedural complications) | 0 | 1
procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 3
pleural effusion (Injury, poisoning and procedural complications) | 0 | 1
respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
chest pain (General disorders) | 2 | 2
fatigue (General disorders) | 0 | 2
headache (Nervous system disorders) | 0 | 2
convulsion (Nervous system disorders) | 1 | 1
cerebrovascular accident (Nervous system disorders) | 1 | 0
tremor (Nervous system disorders) | 0 | 1
depression (Psychiatric disorders) | 0 | 1
mental status change (Psychiatric disorders) | 2 | 0
suicide attempt (Psychiatric disorders) | 0 | 1
calculus urinary (Renal and urinary disorders) | 1 | 0
renal colic (Renal and urinary disorders) | 0 | 1
renal failure (Renal and urinary disorders) | 0 | 1
anaemia (Blood and lymphatic system disorders) | 1 | 1
hyperparathyroidism (Endocrine disorders) | 0 | 1
cholecystitis acute (Hepatobiliary disorders) | 0 | 1
flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=123) | Epoetin Alfa (N=129)
oedema peripheral (General disorders) | 9 | 8
diarrhoea (Gastrointestinal disorders) | 5 | 8
face oedema (General disorders) | 6 | 7
breath sounds abnormal (Respiratory, thoracic and mediastinal disorders) | 4 | 7
pain in extremity (General disorders) | 4 | 7
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 7
back pain (General disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights